CLINICAL TRIAL: NCT00497419
Title: Evaluation of a Fast Track for Patients With STEMI
Brief Title: Reperfusion Time in ST Segment Elevation Myocardial Infarction (STEMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06199
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Myocardial Infarction
Keywords: STEMI; ST elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: fast track

SUMMARY:
Reperfusion delay in STEMI has been shown to be excessive in our community. In order to improve delay a fast track (direct transfer in catheterization laboratory) has been implemented. The present study aims at evaluating the benefits of this procedure.

DETAILED DESCRIPTION:
Reperfusion delay in STEMI has been shown to be excessive in our community. Admission in emergency room and waiting for transfer to catheterization laboratory seems to be the principal source of delay. In order to improve delays a fast track (direct transfer in catheterization laboratory) has been implemented for patients being diagnosed with STEMI by emergency physician out of hospital. The present study aims at evaluating the benefits of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of STEMI

Exclusion Criteria:

* On site resuscitated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Door to balloon time | one year

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Grosgurin, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Emergency Service, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Grosgurin O, Plojoux J, Keller PF, Niquille M, N'koulou R, Mach F, Sarasin FP, Rutschmann OT. Prehospital emergency physician activation of interventional cardiology team reduces door-to-balloon time in ST-elevation myocardial infarction. Swiss Med Wkly. 2010 Apr 17;140(15-16):228-32. doi: 10.4414/smw.2010.12927. PMID 20131111